CLINICAL TRIAL: NCT05930262
Title: Acupuncture Therapy Combined With Breathing Training for Patients With Stroke Complicated With Pulmonary Infection: A Clinical Study
Brief Title: Acupuncture Therapy Combined With Breathing Training for Patients With Stroke Complicated
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, WangHonglian, Principal Investigator, The Second Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ACS002
Record Dates: First submitted 2023-06-06; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Stroke; Lung Diseases
Keywords: Acupuncture therapy; Respiratory training; Seroinflammatory factors; Lung function
MeSH Terms: conditions — Stroke; Lung Diseases | interventions — Rehabilitation; Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Experimental): TCM acupuncture therapy Conventional drug therapy Rehabilitation therapy Breathing training
  Interventions: Device: TCM acupuncture therapy; Drug: Conventional drug therapy; Behavioral: Rehabilitation therapy; Behavioral: Breathing training
- the control group (Active Comparator): Conventional drug therapy Rehabilitation therapy Breathing training
  Interventions: Drug: Conventional drug therapy; Behavioral: Rehabilitation therapy; Behavioral: Breathing training

INTERVENTIONS:
Device: TCM acupuncture therapy — TCM acupuncture therapy: Zusanli, Quchi, Hegu, Taichong, Feishu and Fenglong were selected as the main acupoints, and the auxiliary acupoints were selected according to the symptoms, including Fengchi, Dazhui, Lieque, Tiantu, Shenshu, Zhongfu, etc.
  Arms: the intervention group
Drug: Conventional drug therapy — Antibiotics were selected based on drug sensitivity test results. Patients with body temperature > 38.5℃ were treated with physical cooling and antipyretic drugs. In patients whose sputum was thick and difficult to cough up, nebulization and inhalation therapy was given, as well as effective coughing and patting the back to expel phlegm were guided.
Behavioral: Rehabilitation therapy — Comprehensive training for hemiplegic limbs included a joint range of motion training, bridging exercise, turnover training, balance training, gait training, hand function training and self-care ability training, 40 min/d, 6 times/w.
Behavioral: Breathing training — Training was conducted daily in the morning, or after symptom relief in the case of fever or other discomforts, once a day, 30-40 min/time.

SUMMARY:
The goal of this prospective randomized controlled study is to explore the clinical efficacy of acupuncture therapy combined with breathing training in patients with stroke complicated with pulmonary infection. The intervention group and control group were treated with conventional drug therapy, rehabilitation therapy and breathing training for 2 consecutive weeks. On this basis, the intervention group additionally received acupuncture therapy. To evaluate the clinical efficacy of both groups.

DETAILED DESCRIPTION:
To explore the clinical efficacy of acupuncture therapy combined with breathing training in patients with stroke complicated with pulmonary infection. Using a prospective randomized controlled study, 72 patients with pulmonary infection after stroke admitted to our hospital from May 2020 to May 2021 were randomly divided into the intervention group and control group, with 36 patients in each group. Both groups were treated with conventional drug therapy, rehabilitation therapy and breathing training for 2 consecutive weeks. On this basis, the intervention group additionally received acupuncture therapy. The traditional Chinese medicine (TCM) syndrome score and clinical pulmonary infection score (CPIS) before and after treatment, time of fever relieving, time for the disappearance of cough, expectoration and moist rales in the lung, white blood cell count (WBC), serum C-reactive protein (CRP) level, calcitonin (PCT) level and pulmonary indexes were compared between the 2 groups, respectively, to evaluate clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria of Western medicine for stroke complicated with pneumonia
* conforming to the TCM syndrome of vital qi deficiency and phlegm-heat obstructing the lung
* confirmed as the initial onset of stroke through CT or magnetic resonance imaging (MRI)
* clear consciousness, no cognitive impairment, and ability to cooperate with pulmonary function assessment and rehabilitation training
* willingness to participate in this study and sign the informed consent

Exclusion Criteria:

* Patients with systemic multi-organ failure such as the heart, brain, kidney, etc
* patients with a coronary metal stent or pacemaker implantation
* patients with malignant tumors
* patients with severe cognitive impairment, depression or mental disorders
* patients with pulmonary infections before stroke or caused by other causes
* patients in the acute phase of infection

Ages: 28 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Serum inflammatory factors：C-reactive protein (CRP) level | 2 Weeks
  C-reactive protein (CRP) level(mg/L)
Serum inflammatory factors：Calcitonin (PCT) level | 2 Weeks
  Calcitonin (PCT) level(ng/mL)
Serum inflammatory factors：WBC | 2 Weeks
  WBC (x 109/L)
Improvement time for symptoms and signs of pulmonary infection：Time of fever relieving | 2 Weeks
  the time for body temperature to return to normal (d)
Improvement time for symptoms and signs of pulmonary infection：Time for the disappearance of cough | 2 Weeks
  the time for the disappearance of cough (d)
Improvement time for symptoms and signs of pulmonary infection：Time for the disappearance of expectoration | 2 Weeks
  the time for the disappearance of expectoration (d)
Improvement time for symptoms and signs of pulmonary infection：Time for the disappearance of moist rales | 2 Weeks
  the time for the disappearance of moist rales (d)
TCM syndrome score | 2 Weeks
  Before and after treatment, TCM syndrome scores were counted in the two groups. The main and secondary symptoms were classified into 4 levels, with scores of 0, 1, 2 and 3 based on the severity of the symptoms. The tongue coating and pulse pattern were scored into 2 levels, with no scored as 0 and yes as 1. The sum of various scores was calculated as the total score, with a score range of 0-36. The higher the score, the severer the condition.
Clinical pulmonary infection score (CPIS) | 2 Weeks
  Before and after treatment, the 2 groups were scored comprehensively based on the average range of 12-h body temperature, WBC range, amount and character of tracheal secretions, index of gas exchange, pulmonary infiltration shadow of X-ray chest film, and pathogenic bacteria in sputum culture. According to the severity, they were divided into 3 levels, with a score of 0, 1 and 2. The maximum score was 12. The higher the score, the severer the infection.
Pulmonary indexes:forced vital capacity (FVC) | 2 Weeks
  To measure the forced vital capacity (FVC)(L) before and after treatment
Pulmonary indexes:forced expiratory volume in the first second (FEV1) | 2 Weeks
  To measure the forced expiratory volume in the first second (FEV1)(L/S) before and after treatment
Pulmonary indexes: peak expiratory flow (PEF) | 2 Weeks
  To measure the peak expiratory flow (PEF)(L/S) before and after treatment
Efficacy evaluation:Number of patients with clinical efficacy（Cured，Effective，Remarkably effective，Invalid） | 2 Weeks
  Efficacy was evaluated according to the Criteria of Diagnosis and Therapeutic Effect of Diseases and Symptoms in Traditional Chinese Medicine . Cured: Clinical adverse symptoms such as cough, expectoration and chest tightness disappeared, inflammation was absorbed on X-ray or CT, and routine blood indexes were normal. Remarkably effective: Adverse symptoms such as cough, expectoration and chest tightness were improved significantly, and X-ray or CT and routine blood test results basically returned to normal. Effective: Clinical adverse symptoms such as cough, expectoration and chest tightness were relieved, and X-ray or CT and routine blood test results were improved partially. Invalid: Clinical adverse symptoms such as cough, expectoration and chest tightness had no changes or aggravated.

CONTACTS AND LOCATIONS:
Locations (1):
- Acupuncture Therapy Combined with Breathing Training for Patients with Stroke Complicated with Pulmonary Infection: A Clinical Study, Shijiazhuang, Hebei, China